CLINICAL TRIAL: NCT02638155
Title: Food Addition and Hormone Study
Brief Title: Food Addiction and Hormone Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Cynthia Dsauza, Assistant Professor, Texas Tech University
Other Study IDs: 505490
Record Dates: First submitted 2015-12-03; First posted 2015-12-23 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Disordered Eating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Food Addiction Group: Those participants identified as having food addiction by the Yale Food Addiction Scale.
- No Food Addiction Group: Those participants with no identified food addiction

SUMMARY:
The purpose of this exploratory study is to use Electrogastrography (EGG) to measure and compare the gastric myoelectrical activity between persons with food addiction (FA) and a control group. Additionally, this study will explore if differences exist between perceived hunger and satiety and hormone levels related to hunger and satiety in both groups. The comparison of the EGG readings and hormone levels is the next step in furthering our understanding of food addiction and how the physiology - not simply the symptomatology - of FA does or does not relate to weight management.

DETAILED DESCRIPTION:
The study will be conducted over 2 days and will consist of psychological assessments as well as EGG measurement (similar to EGG) and blood draws to examine hunger and satiety hormones.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include men and women who identify with weight struggles related to disordered eating and a control sample of people who do not identify with weight issues or disordered eating. Must be able to read and write English

Exclusion Criteria:

* Anyone with a chronic disease including type II diabetes, hypothyroidism, hypoparathyroidism, cardiovascular disease, cancer of any type
* Anyone who is currently pregnant, or lactating
* Medications that may influence or inhibit appetite, sensory functioning, or hormone signaling- e.g. antibiotics, anti-depressants, obesity medications
* Report of medical condition or surgical intervention that affects swallowing ability
* Allergy, aversion, or dislike to any of the meal replacements or snacks offered
* Previous or current diagnosis of a psychiatric illness such as schizophrenia or any other psychotic disorder listed in the DSM-IV or DSM-5
* Report of medical conditions that prohibits overnight fasting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men and women 18-65 who are able to come to TTU for testing and meet eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Electrogastrography (EGG) using Bipoac Systems EGG machine | the participant will be tested continuously for approximately 3 1/2 hours on 1 day, readings are collected on a PC
  Skin electrode similar to EKG attached to abdomen and readings taken

SECONDARY OUTCOMES:
Ghrelin | collected via IV catheter over approximately 3 1/2 hours on one day
  hormone assay
Peptide YY | collected via IV catheter over approximately 3 1/2 hours on one day
  hormone assay
GLP-1 | collected via IV catheter over approximately 3 1/2 hours on one day
  hormone assay
Insulin | collected via IV catheter over approximately 3 1/2 hours on one day
  hormone assay
Glucose | collected via IV catheter over approximately 3 1/2 hours on one day
  Blood glucose levels
The Center for Epidemiologic Studies Depression Scale | Day 1-5-10 minutes
  Depression will be measured using The Center for Epidemiologic Studies Depression Scale Revised , a 20-item measure of depression that measures nine different symptom groups of depression according to the American Psychiatric Association Diagnostic and Statistical Manual, fourth edition. These symptom groups include Sadness, Loss of Interest, Appetite, Sleep, Thinking/Concentration, Guilt, Tired, Movement, and Suicidal Ideation. Responses regard frequency of symptoms and are given on 5-point Likert-type scale ranging from 0 (Not at all or less than one day) to 4 (Nearly every day for two weeks). Sample items include "My appetite was poor" and "Nothing made me happy." Item responses are summed to calculate a total score of depression that can be used to classify depression severity. This assessment will take approximately 5-10 minutes.
GAD-7 | Day 1 5-10 minutes
  Anxiety will be measured using the GAD-7 measure used to assess for generalized anxiety disorder and will take less than 5 minutes to complete. The GAD-7 measures anxiety using seven items to assess frequency of anxiety symptoms on which responses are given on a 4-point Likert-type scale ranging from 0 (Not at all) to 3 (Nearly every day). Sample items include "Feeling anxious, nervous, or on edge" and "Becoming easily annoyed or irritable." All items are summed; and higher scores represent higher levels of anxiety and can be used to classify anxiety severity.
Yale Food Addiction Scale 2.0 | Day 1 5-10 minutes
  The YFAS is a 35-item measure developed to operationalize food addiction by assessing signs of substance-dependence symptoms (e.g., tolerance, withdrawal, loss of control) in eating behavior. The YFAS has shown internal consistency, as well as convergent and incremental validity. The YFAS provides 2 scoring options: a symptom count version and a diagnostic version. To receive a "diagnosis" of FA, it is necessary to report experiencing 3 or more symptoms in the past year and clinically significant impairment or distress. The version of the YFAS used in the current study will measure all items on a Likert scale. In line with YFAS scoring instructions, 5 of the Likert scale items were dichotomized, such that participants who indicated that they had never experienced the symptom were assigned a value of zero, and those reporting ever experiencing the symptom in the past year were assigned a value of 1.
Power of Food Scale | Day 1 5-10 minutes
  The Power of Food Scale (PFS) is a 15-item questionnaire on a 5-point Likert scale ranging from 1 (don't agree) to 5 (strongly agree), and it is designed to measure appetite drive towards highly palatable foods through examining appetite-related thoughts, feelings, and motivations
Multidimensional Body-Self Relations Questionnaire - Appearance Scales | Day 1 5-10 minutes
  The Multidimensional Body-Self Relations Questionnaire - Appearance Scales (MBSRQ-AS) is a 34 item measure on a five point Likert scale that is made up of five subscales: Appearance Evaluation, Appearance Orientation, Overweight Preoccupation, Self-Classified Weight, and the Body Areas Satisfaction Scale.
Trait and State Food Cravings Questionnaires | Day 1 5-10 minutes
  The Trait and State Food Cravings Questionnaire is comprised of two questionnaires that measure state (FCQ-S) and trait (FCQ-T) of food cravings. The FCQ-S is comprised of 15 items, and the FCQ-T is comprised of 21 items.
Food Preoccupation Questionnaire | Day 1 5-10 minutes
  The Food Preoccupation Questionnaire (FPQ) is a 26 Likert item questionnaire that measures the frequency and emotionality of thoughts related to food. It is comprised of four subscales: thought frequency as well as positive, negative, and neutral emotional valences.
Automated Self-Administered (ASA) 24 Hour Recall | Day 1 5-10 minutes
  The Automated Self-Administered 24 hour Dietary Recall is a web-based tool that enables automated self-administered 24-hour recalls. It was developed by the National Cancer Institute and has been used in over 200 research studies with over 45,000 participants. Response data are secured at the hosting site using industry standard security controls, including firewalls and encryption.
Resting Metabolic Rate | 10 min
  participant breathes into mouthpiece of handheld device for 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Dsauza, PhD, Principal Investigator — Assistant Professor
Locations (1):
- TTU College of Human Sciences, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No